CLINICAL TRIAL: NCT03038360
Title: CardioSAVE: A 12-months Prospective Longitudinal Controlled Study for the Validation of a Novel Predictive Model and a Diagnostic Tool, for the Risk Stratification of AMI Patients Undergoing PCI
Brief Title: Prospective Study With AMI Patients Undergoing PCI
Acronym: CardioSAVE
Status: Completed | Type: Observational
Sponsor: Firalis SA (Industry)
Collaborators: Herz-Zentrums Bad Krozingen (Other)
Responsible Party: Sponsor
Other Study IDs: ST0033
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CardioSAVE is a prospective 12-month controlled longitudinal study for the validation of a novel predictive model and a diagnostic tool, for the risk stratification of AMI patients undergoing PCI, with a one year follow-up.

DETAILED DESCRIPTION:
Study rational:

Acute Myocardial Infarction (AMI), a common manifestation of coronary artery disease (CAD), is associated with a relatively high incidence and fatality rate. Myocardial Infarction (MI), commonly known as "heart attack", which usually results from an impaired blood supply often caused by thrombus formation in a coronary vessel, resulting in an acute reduction of oxygen supply to a portion of the myocardium. Reperfusion using primary angioplasty through percutaneous coronary intervention (PCI) was proven to be superior to other methods in reducing the fatality rate of the acute phase of the AMI.

During the last decade tremendous efforts have been given to the identification of cardiac biomarkers (BMs) for the diagnosis of AMI. Cardiac BMs have been proven extremely useful in facilitating the diagnostic as well as the timing of therapeutic intervention and in addressing important questions in terms of physiopathology . This resulted in the extensive use of BMs such as troponins in the diagnosis of MI.

Firalis and the Luxembourg general hospital have identified novel biomarkers that could serve as independent risk predictors and prognostic markers for cardiac and clinical complications. First to confirm the value of our identified biomarker panels and to increase their diagnostic/predictive performance, Firalis will identify novel BMs in patient undergoing PCI to include novel biomarkers in this panel and develop a novel early stage prognostic test for clinical outcome in acute myocardial infarction (AMI) patients receiving percutaneous coronary intervention (PCI). This novel test will also be able to monitor treatment response.

For this purpose, the predictive and diagnostic value of the candidate biomarker set have to be clinically validated in a controlled prospective study conducted by the Bad Krozingen Hearth Center. The sample and data collected in this proof of concept study will constitute an independent validation set at the Bad Krozingen Heart Center. Early time point samples will be used to estimate the risk associated with patients and the data obtained will be correlated with the one year outcome of patients.

The development and successful implementation of such diagnostic assay will have strong impact on the quality of care AMI patients, and will significantly reduce costs for healthcare and economy.

Primary objectives:

* To monitor clinical complications registered following PCI, e.g. death, re-infarction and heart failure
* To perform cardiac measurements including electrocardiogram, and left ventricular ejection fraction (LVEF) by cardiac echography and post-AMI myocardium remodelling by cardiac magnetic resonance (CMR) imaging
* To determine the levels of new and exploratory biomarkers in peripheral blood samples collected before and 1 to 3 days after PCI in patients with MI and to correlate them with clinical outcomes.
* To assess the prognostic and diagnostic values of each biomarker or combination of biomarkers prior and shortly (3 and 5 days) after PCI treatment long-term (12 months) clinical outcomes.

Secondary objectives:

* To quantitatively measure reference biomarkers related to cardiac function, including Troponin I/T, CK, CK-MB, BNP, NT-proBNP.
* To correlate the levels of new and exploratory biomarkers with reference biomarkers (Troponin I/T, CK, CK-MB, NT-Pro BNP) and cardiac measurements including electrocardiogram, post-AMI myocardium remodelling by magnetic resonance imaging, and left ventricular ejection fraction (LVEF) by cardiac echography.
* To evaluate the prognostic and diagnostic values of each biomarker or combination with regard to reference biomarkers (Troponin I/T, CK, CK-MB, NT-Pro BNP) as well as the combination of new and reference biomarkers against classical reference biomarkers, and cardiac measurements including regression of ST-segment by electrocardiogram, post-AMI myocardium remodelling by magnetic resonance imaging, and left ventricular ejection fraction (LVEF) by cardiac echography.

Study design:

CardioSAVE is a prospective 12-month controlled longitudinal study in 600 AMI patients, with a one year follow-up conducted by the Bad Krozingen Heart Center. The objectif is to validate a novel predictive model and a diagnostic tool, for the risk stratification of AMI patients undergoing PCI. The sample and data collected by eCRF will allow to set up a prototype personalized medicine device focusing on Heart Failure (HF) induced by AMI. The primary endpoint will be the proportion of patients with left ventricular ejection fraction (LVEF) < 40% at 6 months. The main secondary endpoint is recovery of regional wall motion measured by cMRI at 6 months. Early time point samples, cMRI at day 3 and other clinical patient data will be used to estimate the risk associated with patients and the data obtained will be correlated with the one year outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female patients with non childbearing potential (post-menopausal, ovariectomised or hysterectomised) patients. Menopause is defined as > 60 years, or between 45 and 60 years being amenorrheic for at least 2 years
2. Age more than 18 years old
3. Acute myocardial infarction with clinical decision to treat with percutaneous coronary intervention

   Primary PCI for myocardial infarction:
   * ST-elevation myocardial infarction (STEMI) or
   * Large non-ST-elevation myocardial infarction (NSTEMI) with hs-Troponin T ≥ 0,1 ng/mL
4. Having signed an Informed Consent to participate in the trial before any study related procedure has been taken.
5. Having signed an Informed Consent for Biobank sampling.

Exclusion Criteria:

1. Cardiac arrest, ventricular fibrillation, cardiogenic shock, stent thrombosis, previous AMI, angina within 48h before infarction, previous CABG 3. Severe concomitant non-cardiac illnesses 4. Relevant non-coronary cardiac illnesses 5. Planned major surgery 6. Participated in any investigational drug or therapy study with a non-approved medication, within the previous 3 months 7. Being - dependent on the Investigator or the Sponsor (e.g., including but not limited to affiliated employee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Myocardial Infarction (AMI) patients undergoing Percutaneous Coronary Intervention (PCI)
Sampling Method: Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) < 40% | At 6 months after PCI
  Proportion of patients with LV-EF < 40% at 6 months or Death and/or occurence of serious cardiovascular events such as reinfarction, onset of a cardiovascular disease (e.g. heart failure).

SECONDARY OUTCOMES:
Recovery of regional wall motion | At 6 months after PCI
  Recovery of regional wall motion measured by cMRI at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hueseyin Firat, MD, PhD, Principal Investigator — Firalis SA
Locations (1):
- Universitaets Herz Zentrum, Bad Krozingen, Germany

IPD SHARING:
Plan to Share IPD: No